CLINICAL TRIAL: NCT05586971
Title: A Randomized, Multi-regional, Double-blind, Double-dummy Parallel-group, Placebo and Allopurinol-controlled Phase 3 Study to Assess the Efficacy and Safety of Tigulixostat in Gout Patients With Hyperuricemia
Brief Title: Tigulixostat, Phase 3 Study, Allopurinol Controlled in Gout Patients
Acronym: EURELIA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LG-GDCL010
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Gout; Hyperuricemia; Gout Flare; Tophi
Keywords: Gout; Hyperuricemia; Xanthine Oxidase Inhibitor
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Tigulixostat 100mg (Experimental): Tigulixostat 100mg, Once a day (QD) for up to 12 months
  Interventions: Drug: Tigulixostat
- Tigulixostat 200mg (Experimental): Tigulixostat 200mg, Once a day (QD) for up to 12 months
  Interventions: Drug: Tigulixostat
- Tigulixostat 300mg (Experimental): Tigulixostat 300mg (100mg + 200mg), Once a day (QD) for up to 12 months
  Interventions: Drug: Tigulixostat
- Titrated allopurinol (100-800mg) (Active Comparator): Allopurinol 100-800mg, three times a day (TID) for up to 12 months. The allopurinol dose will be increased in 100 mg increments up to 800mg.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Placebo, three times a day (TID) for up to 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tigulixostat — Xanthine Oxidase Inhibitor
  Other Names: LC350189
  Arms: Tigulixostat 100mg; Tigulixostat 200mg; Tigulixostat 300mg
Drug: Allopurinol — Xanthine Oxidase Inhibitor
  Arms: Titrated allopurinol (100-800mg)
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The aim of this 12-month randomized multi-regional double-blind parallel group allopurinol and placebo-controlled phase 3 study is to assess the efficacy and safety of three different doses of Tigulixostat in gout patients with hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 85 years, inclusive.
* Subjects with hyperuricemia and a history or presence of gout per American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2015 criteria.
* Subjects who are currently on urate-lowering therapies (ULT) with an sUA level ≥6.0 mg/dL at screening (Visit 1); or subjects who are currently not on ULT with an sUA level ≥7.0 mg/dL at screening (Visit 1). Subjects currently on ULT will undergo washout and must have an sUA level ≥7.0 mg/dL at Visit 3 to be randomized and participate in the study.
* Subjects with a Body Mass Index ≤50 kg/m2 and estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 at screening (Visit 1).

Exclusion Criteria:

* Subjects with secondary hyperuricemia and enzymatic defects.
* Subjects experiencing an acute gout attack (intense pain, swelling, or/and tenderness in the joint area) within 2 weeks prior to screening (Visit 1).
* Subjects who have received pegloticase to treat gout which has not responded to the usual treatments.
* Subjects who have not been receiving stable doses of drugs known to affect sUA levels for the last 3 weeks prior to screening (Visit 1).
* Subjects with a history of xanthinuria (elevated levels of xanthine in the urine).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2202 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with sUA levels <6.0 mg/dL sustained at months 4, 5, and 6 | Up to Month 6
  Serum uric acid (sUA) level will be measured at Month 4,5, and 6

SECONDARY OUTCOMES:
The proportion of subjects with sUA levels <5.0 mg/dL sustained at months 4, 5, and 6 | Up to Month 6
  Serum uric acid (sUA) level will be measured at Month 4,5, and 6
Proportion of subjects with at least one gout flare from Month 6 to Month 12. | From Month 6 to Month 12
  Gout flare (intense pain, swelling, or/and tenderness in the joint area) will be assessed from baseline up to 12 months
Proportion of subjects with complete resolution of ≥1 target tophus by Month 12 | Up to Month 12
  Tophi will be measured by independent central blind reader
Incidence rate of adverse event | Up to Month 12
  Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Hyungjin Cho, MD, Study Director — LG Chem
Locations (278):
- United States (123):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alliance for Multispecialty Research, LLC, Daphne, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Syed Research Consultants, LLC, Muscle Shoals, Alabama
  - Syed Research Consultants, LLC, Sheffield, Alabama
  - Arizona Research Clinic, PLLC, Chandler, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Flagstaff, Arizona
  - Arizona Arthritis and Rheumatology Research PLLC, Glendale, Arizona
  - Arizon Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Desert Clinical Research/CCT Research, Mesa, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Fiel Family and Sports Medicine/CCT Research, Tempe, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Velocity Clinical Research, Banning, California
  - American Clinical Trials, Buena Park, California
  - Shreenath Clinical Service, Lakewood, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - TriWest Research Associates, San Diego, California
  - Rheumatology Center of San Diego, San Diego, California
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Herco Medical and Research Center, Inc, Coral Gables, Florida
  - Nouvelle Clinical Research LLC, Cutler Bay, Florida
  - Omega Research Debary, LLC, DeBary, Florida
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Best Quality Research, Inc, Hialeah, Florida
  - New Generation Of Medical Research, LLC, Hialeah, Florida
  - Vital Pharma Research, Hialeah, Florida
  - Accel Research Sites - Lakeland, Lake Mary, Florida
  - Accel Research Sites - St. Petersburg- Largo, Lake Mary, Florida
  - ARS-Matiland Clinical Research Unit, Lake Mary, Florida
  - Homestead Associates in Research,Inc, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - D&H National Research Centers, Inc., Miami, Florida
  - Ivetmar Medical Group, LLC, Miami, Florida
  - Care Research Center Inc, Miami, Florida
  - Pharmax Research of South Florida, Inc, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Miami, Florida
  - M&A Medical Centers and Research, Miami, Florida
  - HMD Research LLC, Orlando, Florida
  - IMA Clinical Research, St. Petersburg, Florida
  - Adult Medicine of Lake County, Inc., Tampa, Florida
  - Research Institute of South Florida, Inc., Tampa, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - Nodal Medical Center, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Clinical Site Partners LLC dba CSP Orlando, Winter Park, Florida
  - Conquest Research, Winter Park, Florida
  - Centricity Research, Columbus, Georgia
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - Vista Clinical Research, LLC, Newnan, Georgia
  - East West Medical Research Institute, Honolulu, Hawaii
  - Family Care Research, LLC, Boise, Idaho
  - Alliance for Multispecialty Research, LLC, Meridian, Idaho
  - IMA Research, Inc., Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - American Health Network of Indiana, LLC, Franklin, Indiana
  - American Health Network of Indiana LLC, Muncie, Indiana
  - Integrated Clinical Trial Services Inc., West Des Moines, Iowa
  - Women's & Family Care LLC, dba GTC Research, Shawnee Mission, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Versailles Family Medicine, Versailles, Kentucky
  - Clinical Trials Management, LLC, Covington, Louisiana
  - Clinical Trials Management, Metairie, Louisiana
  - MD Medical Research, Oxon Hill, Maryland
  - Elite Clinical Research, LLC, Jackson, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Practice Dr David Headley, Port Gibson, Mississippi
  - Healthcare Research Network, Hazelwood, Missouri
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Clay-Platte Family Medicine Clinic, Kansas City, Missouri
  - IMA Clinical Research, St Louis, Missouri
  - St. Louis Medical Professionals, LLC, St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Methodist Physicians Clinic/CCT Research, Fremont, Nebraska
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Healor Primary Care /CCT Research, Las Vegas, Nevada
  - Wake Research - CRCN, Las Vegas, Nevada
  - Alliance for Multispecialty Research, LLC., Las Vegas, Nevada
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - Inspire Santa Fe Medical Group, Santa Fe, New Mexico
  - Long Island Regional Arthritis & Osteoporosis Care PC, Babylon, New York
  - IMA Clinical Research, New York, New York
  - Conquest Research, Vestal, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Triad Clinical Trials, LLC, Greensboro, North Carolina
  - Olympus Family Medicine, Hendersonville, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Carolina Research Center, Inc., Shelby, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Trinity Health Center Medical Arts, Minot, North Dakota
  - Arthritis Associates of Northwest Ohio Inc., Perrysburg, Ohio
  - STAT Research, Vandalia, Ohio
  - Hatboro Medical Associates, P.C., Hatboro, Pennsylvania
  - Tristar Clinical Investigations, P.C., Philadelphia, Pennsylvania
  - New Phase Research, Knoxville, Tennessee
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Inquest Clinical Research, Baytown, Texas
  - PCCR Solutions, Colleyville, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - DFW Clinical Research, Dallas, Texas
  - Dallas Fort Worth Clinical Research Associates, Fort Worth, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - AIM Trials, LLC, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Sugar Lakes Family Practice, PA, Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas
  - Cope Family Medicine/CCT Research, Bountiful, Utah
  - Olympus Family Medicine, Salt Lake City, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - South Ogden Family Medicine Clinic, South Ogden, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Meridian Clinical Research, LLC, Portsmouth, Virginia
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Arthritis Northwest, PLLC, Spokane, Washington
- Argentina (12):
  - Hospital Universitario Austral, Buenos Aires
  - Instituto de Investigaciones Clinicas San Nicolás, Buenos Aires
  - Centro Médico Reumatologico - Organizacion Medica de Investigacion S.A. (OMI), Buenos Aires
  - Aprillus Asistencia e Investigacion Clinica, Buenos Aires
  - Centro Privado de Medicina Familiar, Buenos Aires
  - Clinica Adventista Belgrano, Buenos Aires
  - Instituto de Investigaciones Clinicas Cordoba, Córdoba
  - Centro Integral De Dianogostico por Imagenes Marchegiani (CIDIM), Córdoba
  - Instituto Reumatologico Strusberg, Córdoba
  - Clinica Privada Velez Sarsfield (CPVS), Córdoba
  - Centro de Investigaciones Médicas Tucuman, San Miguel de Tucumán
  - Instituto CAICI (Instituto Centralizado de Asistencia e Investigacion Clinica Integral), Santa Fe
- Australia (5):
  - Emeritus Research (Melbourne), Camberwell
  - Holdsworth House Medical Practice, Darlinghurst
  - Griffith University Clinical Trial Unit, Southport
  - Emeritus Research (Sydney), Sydney
  - The Queen Elizabeth Hospital, Woodville South
- Belgium (3):
  - ReumaClinic, Genk
  - CHU de Liège, Liège
  - CHU HELORA - Hôpital de Mons - Site Kenedy, Mons
- Brazil (8):
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte
  - CETI - Centro de Estudos em Terapias Inovadoras, Curitiba
  - EDUMED - Educação em Saúde S/S Ltda, Curitiba
  - LMK Serviços Médicos Sociedade Simples, Curitiba
  - CMIP-Centro Mineiro de Pesquisa, Juiz de Fora
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - SER - Serviços Especializados em Reumatologia da Bahia, Salvador
  - Clinica Medica Bonfiflioli Ltda, São Paulo
- Bulgaria (8):
  - University Multiprofile Hospital for Active Treatment Plovdiv "Eurohospital" Ltd, Plovdiv
  - Mbal Lyulin EAD, Sofia
  - Medical Center Excelsior OOD, Sofia
  - DCC Fokus-5 Lzip OOD, Sofia
  - Medical Center-N.I. Pirogov EOOD, Sofia
  - Military medical academy, Sofia
  - Acibadem City Clinic Diagnostic And Consultation Center Ltd, Sofia
  - Medical Center Synexus Sofia EOOD, Sofia
- Colombia (4):
  - Centro de Investigacion en Reumatología y Especialidades Médicas S.A.S (CIREEM S.A.S), Bogotá
  - Servimed S.A.S., Bucaramanga
  - IPS Medicos Internistas de Caldas SAS, Manizales
  - Healthy Medical Center SAS, Zipaquirá
- Czechia (5):
  - MUDr. Michaela Blahova, revmatologicka ambulance s.r.o., Brno
  - REVMACLINIC s.r.o., Brno
  - L.K.N Arthrocentrum, Hlučín
  - Revmatologicky ustav, New Town
  - MEDICAL PLUS s.r.o., Uherské Hradiště
- France (6):
  - CHU De Bordeaux, Bordeaux
  - Hôpital Saint Philibert, Lomme
  - Hôpital Edourad Herriot, Lyon
  - Hôpital Lapeyronie, Montpellier
  - Centre Hospitalier Regional D'Orleans, Orléans
  - CHU Hôpitaux De Rouen, Rouen
- Georgia (8):
  - "LJ Clinic" LTD, Kutaisi
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - LTD "Israeli-Georgian Medical Research Clinic Helsicore", Tbilisi
  - Cardioclinic - Digomi Medical Center, Tbilisi
  - JSC "Evex Hospitals", Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
  - LTD MediClub Georgia, Tbilisi
  - Multiprofile Clinic Consilium Medula LTD, Tbilisi
- Germany (8):
  - Emovis GmbH, Berlin
  - Gemeinschaftspraxis Dres. T. und N. Jung, Deggingen
  - Klinische Forschung Dresden GmbH, Dresden
  - Medizentrum Essen Borbeck, Essen
  - Velocity Clincial Research Hamburg GmbH, Hamburg
  - Praxis für klinische Studien, Hamburg
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe
  - Klinische Forschung Schwerin GmbH, Schwerin
- Italy (5):
  - Azienda Ospedaliera Nazionale Ss Antonio E Biagio E C Arrigo Alessandria, Alessandria
  - IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan
  - AOU Policlinico Paolo Giaccone, Palermo
  - AUSL di Reggio Emilia, Arcispedale Santa Maria Nuova-IRCCS, Reggio Emilia
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Kaunas City Polyclinic, Dainava Outpatient Clinic, Kaunas
  - Klaipeda University Hospital, Klaipėda
- Malaysia (8):
  - Hospital Selayang, Batu Caves
  - University Malaya Medical Centre, Kuala Lumpur
  - Klinik Kesihatan Kuang Lumpur, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - Klinik Kesihatan Masjid Tanah, Masjid Tanah
  - Hospital Miri, Miri
  - Klinik Kesihatan Kuang, Rawang
  - Hospital Seri Manjung, Seri Manjung
- New Zealand (10):
  - Southern Clinical Trials Totara, Auckland
  - PCRN Silverdale Medical Centre, Auckland
  - Aotearoa Clinical Trials, Auckland
  - Pacific Clinical Research Network (PCRN) Clinical Trials, Christchurch
  - Lakeland Clinical Trials Waikato, Hamilton
  - Waikato Hospital, Hamilton
  - Southern Clinical Trials Tasman, Nelson
  - Pacific Clinical Research Network (PCRN) - Rotorua, Rotorua
  - Lakeland Clinical Trials Wellington, Wellington
  - Wellington Regional Hospital, Wellington
- Philippines (14):
  - Angeles University Foundation Medical Center, Angeles
  - Baguio General Hospital and Medical Center, Baguio City
  - Cebu Doctors' University Hospital, Cebu
  - De la Salle Medical and Health Sciences Institute, Dasmariñas
  - Davao Doctors Hospital, Davao City
  - Iloilo Doctors' Hospital Inc, Iloilo City
  - St. Paul's Hospital of Iloilo, Iloilo City
  - Lipa Medix Medical Center, Lipa
  - Ospital ng Makati, Makati
  - Makati Medical Center, Makati
  - Manila Doctors Hospital, Manila
  - Medical Center Manila, Manila
  - University of the Philippines - Philippine General Hospital, Manila
  - Chinese General Hospital and Medical Center, Manila
- Poland (13):
  - ClinicMed Daniluk, Nowak Spdtka komandytowa, Bialystok
  - Centrum Kliniczno-Badawcze J.Brzezicki, B.Gornikiewicz-Brzezicka Lekarze Spolka Partnerska, Elblag
  - Malopolskie Centrum Kliniczne, Krakow
  - Pratia MCM Krakow, Krakow
  - Centrum Medyczne PROMED, Krakow
  - SOMED CR, Lodz
  - Zespol Poradni Specjalistycznych REUMED, Filia nr 1 Wallenroda, Lublin
  - ETYKA - Ośrodek Badań Klinicznych, Olsztyn
  - FutureMeds Warszawa Centrum, Warsaw
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. prof. dr hab. med. Eleonory Reicher, Warsaw
  - FutureMeds Targéwek, Warsaw
  - Reum-Medica S.C. Bozena Kowalewska, Marek Zawadzki, Wroclaw
- South Korea (9):
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Jeju National University Hospital, Jeju City
  - Kyunghee University Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Uijeongbu Eulji Medical Cen, Uijeongbu-si
- Spain (12):
  - Hospital Universitario de A Coruña, A Coruña
  - HM Hospital Nuestra Señora de la Esperanza, A Coruña
  - Hospital Clinico Universitario de Santiago de Compostela (CHUS), A Coruña
  - Hospital Sanitas CIMA, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Gaias Santiago, Santiago de Compostela
  - Hospital Quirónsalud Sagrado Corazón, Seville
  - Hospital do Meixoeiro, Vigo
- Taiwan (6):
  - Chang Gung Medical Foundation - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - Chang Gung Medical Foundation - Linkou Chang Gung Memorial Hospital, Taoyuan
- Thailand (8):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Thammasat University Hospital, Khlong Luang
  - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saag KG, Dalbeth N, Hsu CY, Kuo CF, Nuki G, Perez-Ruiz F, White WB, Hariri A, Lee Y, Jang Y, Han S, Choi HK. Evaluation of the efficacy and safety of a novel xanthine oxidase inhibitor, tigulixostat, in gout patients with hyperuricemia: Design of the EURELIA 1 and EURELIA 2 studies. Contemp Clin Trials. 2025 Apr;151:107843. doi: 10.1016/j.cct.2025.107843. Epub 2025 Feb 8. PMID 39929260